CLINICAL TRIAL: NCT00869388
Title: A Phase I Study of Bi-Weekly rBBX-01 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-0961
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Solid Tumors
Keywords: malignant; resistant; solid tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental): rBBX-01 1.0 mg/m2 SC on 5 consecutive days on weeks 1, 3, 5, and 7
  Interventions: Biological: rBBX-01
- Arm 2 (Experimental): rBBX-01 2.0 mg/m2 SC on 5 consecutive days on weeks 1, 3, 5, and 7
  Interventions: Biological: rBBX-01
- Arm 3 (Experimental): rBBX-01 4.0 mg/m2 SC on 5 consecutive days on weeks 1, 3, 5, and 7
  Interventions: Biological: rBBX-01
- Arm 4 (optional) (Experimental): rBBX-01 8.0 mg/m2 SC on 5 consecutive days on weeks 1, 3, 5, and 7
  Interventions: Biological: rBBX-01

INTERVENTIONS:
Biological: rBBX-01

SUMMARY:
This study will evaluate toxicity associated with escalating doses of rBBX-01 given bi-weekly to patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed metastatic or unresectable, resistant solid tumor. Gynecologic tumors preferred.
* 18 years and above
* GOG performance status greater than or equal to 2
* Life expectancy greater than 6 months
* Acceptable organ and marrow function
* Willingness to agree to use adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Not receiving any other investigational agents
* Known brain metastasis
* Uncontrolled intercurrent illness including, but not limited to ongoing ore active infection, symptomatic congestive heart failure, unstable angina pectoris,cardiac arrythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy
* Immunosuppression including subjects with known HIV infection on immunosuppressive drugs or having an autoimmune disorder
* Penicillin allergy
* Symptomatic prostate hypertrophy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To determine the dose limiting toxicity and safety of bi-weekly courses of rBBX-01 in patients with resistant solid tumor malignancies. | Four bi-weekly 5 day courses

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic and pharmacodynamics of bi-weekly rBBX-01. To correlate the inter-patient sensitivity to rBBX-01 with in vitro studies on patient blood. To describe any anti-tumor activity of rBBX-01. | 4 bi-weekly 5 day courses

CONTACTS AND LOCATIONS:
Overall Officials: Premal Thaker, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Basche M, Gustafson DL, Holden SN, O'Bryant CL, Gore L, Witta S, Schultz MK, Morrow M, Levin A, Creese BR, Kangas M, Roberts K, Nguyen T, Davis K, Addison RS, Moore JC, Eckhardt SG. A phase I biological and pharmacologic study of the heparanase inhibitor PI-88 in patients with advanced solid tumors. Clin Cancer Res. 2006 Sep 15;12(18):5471-80. doi: 10.1158/1078-0432.CCR-05-2423. PMID 17000682
- [Background] Hayashi N, Kinoshita H, Yukawa E, Higuchi S. Pharmacokinetic and pharmacodynamic analysis of subcutaneous recombinant human granulocyte colony stimulating factor (lenograstim) administration. J Clin Pharmacol. 1999 Jun;39(6):583-92. doi: 10.1177/00912709922008191. PMID 10354962
- [Background] Rosenberg B, Juckett DA, Aylsworth CF, Dimitrov NV, Ho SC, Judge JW, Kessel S, Quensen J, Wong KP, Zlatkin I, Zlatkin T. Protein from intestinal Eimeria protozoan stimulates IL-12 release from dendritic cells, exhibits antitumor properties in vivo and is correlated with low intestinal tumorigenicity. Int J Cancer. 2005 May 1;114(5):756-65. doi: 10.1002/ijc.20801. PMID 15609305
- [Background] Rader JS, Aylsworth CF, Juckett DA, Mutch DG, Powell MA, Lippmann L, Dimitrov NV. Phase I study and preliminary pharmacology of the novel innate immune modulator rBBX-01 in gynecologic cancers. Clin Cancer Res. 2008 May 15;14(10):3089-97. doi: 10.1158/1078-0432.CCR-07-4250. PMID 18483376
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu